CLINICAL TRIAL: NCT00072657
Title: Behavioral Treatments for Rheumatoid Arthritis
Brief Title: Cognitive-Behavioral Therapy and Tai Chi Chih for Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Perry Nicassio, Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AR049840 (NIH); R01AR049840 (NIH); NIAMS-095
Record Dates: First submitted 2003-11-07; First posted 2003-11-10 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis; Pain; Meditation; Tai Chi; Chronic Illness; Depression
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Pain; Chronic Disease; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- 1 (Experimental): Participants will partake in cognitive behavioral therapy for 12 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- 2 (Experimental): Participants will partake in tai chi chih for 12 weeks.
  Interventions: Behavioral: Tai Chi Chih
- 3 (Active Comparator): Participants will act as a control and attend educational sessions for 12 weeks.
  Interventions: Behavioral: Health Education Seminar

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — The CBT intervention will have three phases: 1) education on the nature of the adjustment process in chronic illness, 2) coping skill development, and 3) generalization and application of skills to everyday situations. Participants in the CBT group will attend 12 weekly group sessions of about 2 hours each.
  Arms: 1
Behavioral: Tai Chi Chih — Participants in the TCC group will learn to perform 18 movements under the guidance of an expert TCC teacher. TCC participants will have 50- to 60-minute biweekly sessions during the 12-week study.
  Arms: 2
Behavioral: Health Education Seminar — Control group participants will attend weekly group educational sessions; these sessions will provide general knowledge about arthritis health and illness, and they will include lectures, demonstrations, and question-and-answer sessions with experts in rheumatology, sleep science, and behavioral medicine.
  Arms: 3

SUMMARY:
Rheumatoid arthritis (RA) is a chronic illness. Patients with RA often experience significant pain and depression. This study will evaluate two programs designed to improve the symptoms of RA: cognitive-behavioral therapy (CBT) and Tai Chi Chih (TCC), compared to a health education seminar.

DETAILED DESCRIPTION:
Rheumatoid arthritis is a progressive inflammatory illness marked by severe functional declines, significant economic and social costs, and significant psychological distress. Environmental and psychosocial factors such as stress, mood disturbance, and coping mechanisms may contribute to changes in important health outcomes, including disability and disease activity in RA. This study will compare CBT with TCC, a relaxation-based intervention, combining elements of slow gentle movement with meditation, against a more traditional health education seminar. Outcome measures will include psychological adaptation, mood disturbance, sleep quality, physiological adaptation, and disease severity.

Two hundred-ten patients will be randomly assigned to either CBT, TCC, or a control group. The CBT intervention will have three phases: 1) education on the nature of the adjustment process in chronic illness, 2) coping skill development, and 3) generalization and application of skills to everyday situations. Participants in the CBT group will attend 12 weekly group sessions of about 2 hours each. Participants in the TCC group will learn to perform 18 movements under the guidance of an expert TCC teacher. TCC participants will have 50 to 60 minute biweekly sessions during the 12-week study. Control group participants will attend weekly group educational sessions; these sessions will provide general knowledge about arthritis health and illness, and will include lectures, demonstrations, and question-and-answer sessions with experts in rheumatology, sleep science, and behavioral medicine.

Participants will be assessed prior to beginning treatment, at mid-treatment (Week 6) and again at the end of treatment (Week 12 to 13). The long term effect of interventions will be assessed at follow-up interviews 4 months and 8 months after the end of formal treatment. Psychosocial adaptation, mood disturbance and sleep quality, self-reported pain, and immune function will be measured at all five assessment periods.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA as defined by the American College of Rheumatology (ACR) and consistent with revised criteria for RA
* Stable disease-modifying drug regimen for 3 months prior to study entry, with no change in drug dosage for at least 3 months prior to study entry
* Relatively stable disease course for 3 months prior to study entry
* If treated with corticosteroids, must be on a stable dosage for 3 months prior to study entry
* If taking prednisone, must be on a dosage less than or equal to 10 mg/day or equivalent
* Resides in Greater Los Angeles area

Exclusion Criteria:

* Inactive RA conditions defined as "in remission"
* Experiencing frequent, severe disease flares that require changes in primary disease-modifying regimen
* Serious medical conditions, including: diabetes, congestive heart failure, renal failure requiring specific treatment, cancer (unless cured for period of 5 years or more), unregulated endocrine disorders (including thyroid disorders), chronic uncontrolled infection, or any uncontrolled medical condition that may interfere with the study
* Use of analgesics (e.g., opioids) other than acetaminophen or non-steroidal anti-inflammatory agents prescribed for RA treatment, tramadol (Ultram) or Tylenol with codeine on an as-needed basis, or propoxyphen (Darvocet, Wygesic)
* Use of oxycodone (Percocet), hydrocodone (Vicodin), morphine, or hydromorphone (Dilaudid)
* Use of high levels of methotrexate (greater than 7.5 mg)
* Use of nitrogen mustard, cyclosporine, monoclonal antibodies, or cyclophosphamide within the 6 months prior to study entry
* Serious psychiatric conditions, such as bipolar disorder, psychotic disorders, or organic brain syndromes
* At risk for suicide
* Dependent on canes, walkers, or other assistive devices
* Unable to commit to study schedule/itinerary or unwilling to be assigned to any of the 3 treatment groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2004-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Disease activity | Measured at Week 12 and Months 4 and 8 follow-up
Health functioning | Measured at Week 12 and Months 4 and 8 follow-up
Inflammation, measured by levels of IL-1, IL-6, and tumor necrosis factor (TNF)-alpha | Measured at Week 12 and Months 4 and 8 follow-up

SECONDARY OUTCOMES:
Mood disturbances | Measured at Week 12 and Months 4 and 8 follow-up
Coping | Measured at Week 12 and Months 4 and 8 follow-up
Helplessness | Measured at Week 12 and Months 4 and 8 follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Perry M. Nicassio, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Cousins Center for Psychoneuroimmunology, UCLA, Los Angeles, California, United States

REFERENCES:
- [Derived] Azizoddin DR, Olmstead R, Anderson KA, Hirz AE, Irwin MR, Gholizadeh S, Weisman M, Ishimori M, Wallace D, Nicassio P. Socioeconomic status, reserve capacity, and depressive symptoms predict pain in Rheumatoid Arthritis: an examination of the reserve capacity model. BMC Rheumatol. 2024 Sep 20;8(1):46. doi: 10.1186/s41927-024-00416-4. PMID 39304956
- [Derived] Azizoddin D, Olmstead R, Anderson KA, Hirz AE, Irwin MR, Gholizadeh S, Weisman M, Ishimori M, Wallace D, Nicassio P. Socioeconomic Status, Reserve Capacity, and Depressive Symptoms Predict Pain in Rheumatoid Arthritis: An Examination of the Reserve Capacity Model. Res Sq [Preprint]. 2023 Apr 7:rs.3.rs-2758092. doi: 10.21203/rs.3.rs-2758092/v1. PMID 37066198
- [Derived] Ormseth SR, Draper TL, Irwin MR, Weisman MH, Arechiga AE, Hartoonian N, Bui T, Nicassio PM. Multidimensional Model of Disability and Role Functioning in Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2015 Dec;67(12):1686-92. doi: 10.1002/acr.22658. PMID 26212464